CLINICAL TRIAL: NCT04289584
Title: Efficacy of a Physiotherapy Intervention Through Exercises With Elastic Bands and Stability Exercises in the Improvement of Proprioception and Strength During Unipodal Support in Women Athletes of Taekwondo. A Randomized Clinical Study.
Brief Title: Exercises With Elastic Bands and Stability in Proprioception and Strength in Female Athletes of Taekwondo
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Lockdown
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TKD
Record Dates: First submitted 2020-02-27; First posted 2020-02-28 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Proprioceptive Disorders
Keywords: Taekwondo; Strength; Balance; Theraband; Proprioception
MeSH Terms: conditions — Somatosensory Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Each session will last 15 minutes, taking place for 2 days a week, over a period of 4 weeks. The intervention will take place at the beginning of the training session. Prior to training, strength and proprioception exercises will be performed.
  Interventions: Other: Strength and proprioception exercises
- Control group (No Intervention): The players included in the control group will follow their usual routine prior to their Taekwondo training.

INTERVENTIONS:
Other: Strength and proprioception exercises — Strength and proprioception exercises will be performed with the athlete in different positions depending on the exercise. There will be 3 series with 30 repetitions and 10-second breaks between sets. Each exercise session will be held for 15 minutes. Theraband® exercises are: unipodal balancing on hard surface with open and closed eyes, unipodal balancing on soft surface, squats, lateral walk, isometric contractions with garter and dynamic leg opening, tiptoe, and eccentric hamstring curl with garter.
  Arms: Experimental group

SUMMARY:
Strength and proprioception exercises are used to improve the strength and unipodal balance of lower limbs in Taekwondo players. The moments of unipodal support in Taekwondo require a great demand that is necessary to adapt the athlete through the development of strength and proprioception.

The main objective of the study is to assess the effectiveness of strength work with elastic bands and balance exercises in increasing strength and unipodal proprioception in taekwondists aged 18 to 30 years.

Randomized, single blind clinical study 30 taekwondists will be randomized to the two study groups: experimental (strength training and proprioception) and control (without intervention). The intervention will last 4 weeks, with 2 weekly sessions each session will be approximately 15 minutes each. The study variables will be: unipodal muscle strength (jump test), and lower limb balance (Y-Balance test). The sample distribution will be calculated using a Kolmogorov-Smmirnof analysis. The changes after each evaluation will be analyzed with the t-student test and with an ANOVA of repeated measures the intra and intersubject effect will be observed. The effect size will be calculated using Cohen's formula.

After the training period it is intended to obtain improvement in the strength of the lower limbs, as well as an increase in balance during unipodal support during the execution of a movement.

ELIGIBILITY:
Inclusion Criteria:

* Female Taekwondo players
* Age range of 18 to 30 years
* More than 2 years of sports practice of taekwondo, federated
* Currently participate in regional or national competitions.

Exclusion Criteria:

* Participants who have some type of musculoskeletal lesion in the lower limbs
* That are belts below the color green
* Have not competed in the last year in any regional or national competition.
* Have not signed the informed consent document

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline strength after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be done using the Hop test, measuring the single jump for distance The test will be done twice and the result will be the average of the two values to calculate the symmetry of the limbs. Before carrying out the test it is necessary to create a horizontal line as a starting point and six meters to there a horizontal line as an end point. A vertical 15 cm line will be placed as a reference point for the cross jump from the starting line to the finishing line. The simple jump of distance consists in realizing a jump starting from a monopodal support and falling of the jump with the same leg that realizes the impulse. The unit of measure is the centimeter, based on the distance traveled.

SECONDARY OUTCOMES:
Change from baseline stability after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be done by applying the Y-Balance test. With this test, the unipodal stability of each lower limb will be measured. To perform the test you must create a "Y" figure on the floor. The athlete will place one foot barefoot at the central point of the "Y", while the other foot should be carried along the lines in the 3 directions: anterior, posterolateral and posteromedial. The players will be asked to stretch their foot as much as possible without losing their balance, then returning to the starting point. Three repetitions will be performed and the result will be the average of these measures. There will be a 15 second break between each unilateral take and 30 seconds between each foot.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain